CLINICAL TRIAL: NCT02698475
Title: A Phase 3 Open-label Study to Assess the Efficacy, Safety, and Pharmacokinetics of Subcutaneously Administered Ustekinumab in the Treatment of Moderate to Severe Chronic Plaque Psoriasis in Pediatric Subjects Greater Than or Equal to 6 to Less Than 12 Years of Age
Brief Title: An Efficacy, Safety, and Pharmacokinetics Study of Subcutaneously Administered Ustekinumab in the Treatment of Moderate to Severe Chronic Plaque Psoriasis in Pediatric Participants Greater Than or Equal to 6 to Less Than 12 Years of Age
Acronym: CADMUS Jr
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108129; CNTO1275PSO3013 (Other: Janssen Research & Development, LLC); 2016-000121-40 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Psoriasis
Keywords: Psoriasis; Ustekinumab; STELARA
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ustekinumab Group (Experimental): Participants will receive 1 of the following dose levels depending on their weight: participants weighing less than (<) 60 kg will receive Ustekinumab 0.75 milligram per kilogram (mg/kg); participants weighing greater than or equal to (>=) 60 kg to less than or equal to (<=) 100 kg will receive ustekinumab 45 mg; participants weighing >100 kg will receive ustekinumab 90 mg, at Weeks 0 and 4 followed by every 12 weeks dosing with the last dose at Week 40. Eligible participants who enter the long-term extension (LTE) period will continue receiving ustekinumab every 12 weeks (q12w) beginning at Week 56 up to Week 248.
  Interventions: Drug: Ustekinumab 0.75 mg/kg; Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg

INTERVENTIONS:
Drug: Ustekinumab 0.75 mg/kg — Participants weighing less than (<) 60 kilograms will receive ustekinumab 0.75 milligram per kilogram (mg/kg) at Weeks 0 and 4 followed by every 12 weeks dosing with the last dose at Week 40. Eligible participants for LTE period will continue to receive ustekinumab 0.75 mg/kg up to Week 248.
Drug: Ustekinumab 45 mg — Participants weighing greater than or equal to (>=) 60 kg to less than or equal to (<=) 100 kg will receive ustekinumab 45 mg at Weeks 0 and 4 followed by every 12 weeks dosing with the last dose at Week 40. Eligible participants for LTE period will continue to receive ustekinumab 45 mg up to Week 248.
Drug: Ustekinumab 90 mg — Participants weighing >100 kg will receive ustekinumab 90 mg at Weeks 0 and 4 followed by every 12 weeks dosing with the last dose at Week 40. Eligible participants for LTE period will continue to receive ustekinumab 90 mg up to Week 248.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ustekinumab in pediatric participants aged greater than or equal to (>=) 6 through less than (<) 12 years with moderate to severe chronic plaque psoriasis

DETAILED DESCRIPTION:
This is an open label (identity of study drug will be known to participant and study staff) and multicenter (when more than one hospital or medical school team work on a medical research study) study. The participant population will be comprised of boys and girls who have had a diagnosis of plaque psoriasis for at least 6 months prior to first study drug administration and who have moderate to severe disease defined by Psoriasis Area and Severity Index score (PASI) >=12, Physician's Global Assessment (PGA) >=3, and Body Surface Area (BSA) >=10 percent (%). The study consists of Screening Phase (up to 10 weeks before administration of the study drug), Treatment Period (Week 0 up to Week 52) and Safety follow up (Week 56). Participants will be primarily evaluated for efficacy, pharmacokinetics (PK) and safety. Following completion of the Week 52 visit, participants who have had a beneficial response from ustekinumab treatment as determined by the investigator, and who have not yet reached the age of 12 years or older in countries where marketing authorization for ustekinumab has been granted for the treatment of psoriasis in adolescent participants (12-17 years), and are willing to continue ustekinumab treatment, may enter the long-term extension period (from Week 56 through Week 264) of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have a diagnosis of plaque-type psoriasis with or without psoriatic arthritis (PsA) for at least 6 months prior to first administration of study drug, with widespread lesions defined by Psoriasis Area and Severity Index score (PASI) greater than or equal to (>=) 12, Physician's Global Assessment (PGA) >=3, and involved body surface area (BSA) >=10 percent (%)
* Participants who are candidates for phototherapy or systemic treatment of psoriasis (either naive or history of previous treatment) or have psoriasis considered by the investigator as poorly controlled with topical therapy after an adequate dose and duration of therapy
* Participants who are considered eligible according to the protocol defined tuberculosis (TB) screening criteria
* Participants must have positive protective antibody titers to varicella and measles prior to the first administration of study drug. In the absence of positive protective antibody titers, the participant must have documentation of age-appropriate vaccination for varicella and/or measles (that includes both doses of each vaccine) or verification of past varicella and/or measles infection documented by a health care provider
* Participants must agree not to receive a live virus or live bacterial vaccination at least 2 weeks (or longer as indicated in the package insert of the relevant vaccine) prior to the first administration of study drug, during the study, or within 15 weeks after the last administration of study drug
* Participants must agree not to receive a Bacille Calmette-Guerin (BCG) vaccination within 12 months of screening, during the study, or within 12 months after the last administration of study drug

Exclusion Criteria:

* Participants who currently have nonplaque forms of psoriasis (example, erythrodermic, guttate, or pustular)
* Have received any systemic immunosuppressants (example methotrexate [MTX], azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, and tacrolimus) within 4 weeks of the first administration of study drug
* Have received any biologic agent (example ENBREL, HUMIRA) within the previous 3 months or 5 times the t1/2 of the agent, whichever is longer
* Have a history of chronic or recurrent infectious disease
* Have a history of latent or active granulomatous infection
* Have any known malignancy or have a history of malignancy
* Have a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (31):
- United States (7):
  - San Diego, California
  - Chicago, Illinois
  - Indianapolis, Indiana
  - St Louis, Missouri
  - Arlington, Texas
  - Dallas, Texas
  - Norfolk, Virginia
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Canada (2):
  - Calgary, Alberta
  - St. John's, Newfoundland and Labrador
- Germany (4):
  - Berlin
  - Bonn
  - Dresden
  - Frankfurt
- Hungary (5):
  - Budapest
  - Debrecen
  - Kaposvár
  - Kecskemét
  - Szeged
- Nijmegen, Netherlands
- Poland (3):
  - Lodz
  - Warsaw
  - Wroclaw
- South Korea (3):
  - Bundang
  - Incheon
  - Seoul
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District

REFERENCES:
- [Derived] Leu JH, Shiff NJ, Clark M, Bensley K, Lomax KG, Berezny K, Nelson RM, Zhou H, Xu Z. Intravenous Golimumab in Patients with Polyarticular Juvenile Idiopathic Arthritis and Juvenile Psoriatic Arthritis and Subcutaneous Ustekinumab in Patients with Juvenile Psoriatic Arthritis: Extrapolation of Data from Studies in Adults and Adjacent Pediatric Populations. Paediatr Drugs. 2022 Nov;24(6):699-714. doi: 10.1007/s40272-022-00533-y. Epub 2022 Sep 28. PMID 36171515

RESULTS

PARTICIPANT FLOW:
Groups:
- Ustekinumab Standard Dosage: Participants received ustekinumab standard weight-based dose at Weeks 0 and 4 followed by every 12 weeks (q12w) dosing up to Week 40. Ustekinumab was administered as subcutaneous (SC) injections of 0.75 milligrams per kilogram (mg/kg) for participants with weight less than (<) 60 kilograms (kg), 45 mg for participants with weight greater than or equal to (>=) 60 kg to less than or equal to (<=) 100 kg, and 90 mg for participants with weight > 100 kg. Participants had a safety follow-up till Week 56 (Main study period). During long-term extension (LTE) period, participants who had a beneficial response from ustekinumab treatment continued receiving ustekinumab weight based dose in a q12w regimen from Week 56 onwards until commercially available or marketing authorization being denied or up to Week 264.
Period: Main Study Period
Arm/Group | Ustekinumab Standard Dosage
Started | 44
Completed | 41
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 2
Period: Long-Term Extension Period
Arm/Group | Ustekinumab Standard Dosage
Started | 28 (13 participants did not enter the long-term extension period.)
Completed | 0
Not Completed | 28
Not completed — Lost to Follow-up | 1
Not completed — Trial Site Terminated by Sponsor | 1
Not completed — Withdrawal by Subject | 3
Not completed — Due to Long Term Extension Protocol-Specified Criteria | 22
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ustekinumab Standard Dosage
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 1
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4
  Canada | 2
  Germany | 7
  Hungary | 10
  Netherlands | 1
  Poland | 12
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Physician's Global Assessment (PGA) Score of Cleared (0) or Minimal (1) at Week 12
Description: The PGA is used to determine the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), marked (4), or severe (5). Higher scores indicate worse disease. Treatment Failure (TF) criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Week 12
Population: Full analysis set (FAS): all enrolled and treated participants who received at least 1 injection of ustekinumab (partial or complete). Participants who met TF criteria prior to Week 12 or with missing data at Week 12 were considered non-responders at Week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ustekinumab Standard Dose (Main Study): Participants received ustekinumab -standard weight-based dose at Weeks 0 and 4 followed by q12w dosing up to Week 40. Ustekinumab was administered as SC injections of 0.75 mg/kg for participants with weight <60 kg, 45 mg for participants with weight >=60 kg to <=100 kg, and 90 mg for participants with weight >100 kg. Participants had a safety follow-up till Week 56.
Arm/Group | Ustekinumab Standard Dose (Main Study)
Number analyzed (Participants) | 44
percentage of participants | 77.3 [62.2 to 88.5]

2. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index (PASI) 75 Response at Week 12
Description: PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. Participants with >=75% improvement in PASI from baseline were considered PASI 75 responders. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Week 12
Population: FAS. Participants who met TF criteria prior to Week 12 or with missing data at Week 12 were considered non-responders at Week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ustekinumab Standard Dosage (Main Study): Participants received ustekinumab -standard weight-based dose at Weeks 0 and 4 followed by q12w dosing up to Week 40. Ustekinumab was administered as SC injections of 0.75 mg/kg for participants with weight <60 kg, 45 mg for participants with weight >=60 kg to <=100 kg, and 90 mg for participants with weight >100 kg. Participants had a safety follow-up till Week 56.
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
percentage of participants | 84.1 [69.9 to 93.4]

3. Secondary Outcome: Change From Baseline in Children Dermatology Life Quality Index (CDLQI) Score at Week 12
Description: CDLQI was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (Not at all) to 3 (Very much). The total score ranges from 0 to 30, with lower scores indicating better quality of life. The higher the score, the greater the impairment in quality of life (QoL). TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Baseline and Week 12
Population: FAS. For participants meeting one or more TF criteria, were considered to have 0 improvement from baseline. Here "N" (number of participants analyzed) signifies participants who were evaluable for this outcome measure at both baseline and Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 42
units on a scale | -6.3 (6.43)

4. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Week 12
Description: PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72 (disease severity). A higher score indicates more severe disease. Participants with >=90% improvement in PASI from baseline were considered PASI 90 responders. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
percentage of participants | 63.6 [47.8 to 77.6]

5. Secondary Outcome: Percentage of Participants With a PGA Score of Cleared (0), Cleared (0) or Minimal (1), Mild (2) at Weeks 4, 8, 12, 16, 28, 40, and 52
Description: The PGA is used to determine the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), marked (4), or severe (5). Higher scores indicate worse disease. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Weeks 4, 8, 12, 16, 28, 40, and 52
Population: FAS. Participants who met 1 or more TF criteria were considered as non-responders after TF. In addition, participants with missing data at Week 12 were also considered as non-responders at Week 12. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
percentage of participants
  Week 4: PGA Score 0: number analyzed (Participants) | 42
  Week 4: PGA Score 0 | 4.8
  Week 4: PGA Score 0 or 1: number analyzed (Participants) | 42
  Week 4: PGA Score 0 or 1 | 33.3
  Week 4: PGA Score 0 or 1 or 2: number analyzed (Participants) | 42
  Week 4: PGA Score 0 or 1 or 2 | 66.7
  Week 8: PGA Score 0: number analyzed (Participants) | 41
  Week 8: PGA Score 0 | 26.8
  Week 8: PGA Score 0 or 1: number analyzed (Participants) | 41
  Week 8: PGA Score 0 or 1 | 63.4
  Week 8: PGA Score 0 or 1 or 2: number analyzed (Participants) | 41
  Week 8: PGA Score 0 or 1 or 2 | 85.4
  Week 12: PGA Score 0 | 38.6
  Week 12: PGA Score 0 or 1 | 77.3
  Week 12: PGA Score 0 or 1 or 2 | 90.9
  Week 16: PGA Score 0: number analyzed (Participants) | 42
  Week 16: PGA Score 0 | 45.2
  Week 16: PGA Score 0 or 1: number analyzed (Participants) | 42
  Week 16: PGA Score 0 or 1 | 85.7
  Week 16: PGA Score 0 or 1 or 2: number analyzed (Participants) | 42
  Week 16: PGA Score 0 or 1 or 2 | 95.2
  Week 28: PGA Score 0: number analyzed (Participants) | 42
  Week 28: PGA Score 0 | 45.2
  Week 28: PGA Score 0 or 1: number analyzed (Participants) | 42
  Week 28: PGA Score 0 or 1 | 83.3
  Week 28: PGA Score 0 or 1 or 2: number analyzed (Participants) | 42
  Week 28: PGA Score 0 or 1 or 2 | 95.2
  Week 40: PGA Score 0: number analyzed (Participants) | 42
  Week 40: PGA Score 0 | 52.4
  Week 40: PGA Score 0 or 1: number analyzed (Participants) | 42
  Week 40: PGA Score 0 or 1 | 76.2
  Week 40: PGA Score 0 or 1 or 2: number analyzed (Participants) | 42
  Week 40: PGA Score 0 or 1 or 2 | 90.5
  Week 52: PGA Score 0: number analyzed (Participants) | 41
  Week 52: PGA Score 0 | 56.1
  Week 52: PGA Score 0 or 1: number analyzed (Participants) | 41
  Week 52: PGA Score 0 or 1 | 75.6
  Week 52: PGA Score 0 or 1 or 2: number analyzed (Participants) | 41
  Week 52: PGA Score 0 or 1 or 2 | 90.2

6. Secondary Outcome: Percentage of Participants Who Achieved a PASI 50, PASI 75, PASI 90 and PASI 100 Response at Weeks 4, 8, 12, 16, 28, 40, and 52
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72 (disease severity). PASI 50, 75, 90, and 100 responders were defined as >=50%, >=75%, >=90%, and 100% improvement in PASI from Baseline respectively. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Weeks 4, 8, 12, 16, 28, 40, and 52
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
percentage of participants
  Week 4: PASI 100: number analyzed (Participants) | 42
  Week 4: PASI 100 | 2.4
  Week 4: PASI 90: number analyzed (Participants) | 42
  Week 4: PASI 90 | 16.7
  Week 4: PASI 75: number analyzed (Participants) | 42
  Week 4: PASI 75 | 26.2
  Week 4: PASI 50: number analyzed (Participants) | 42
  Week 4: PASI 50 | 52.4
  Week 8: PASI 100: number analyzed (Participants) | 41
  Week 8: PASI 100 | 17.1
  Week 8: PASI 90: number analyzed (Participants) | 41
  Week 8: PASI 90 | 43.9
  Week 8: PASI 75: number analyzed (Participants) | 41
  Week 8: PASI 75 | 58.5
  Week 8: PASI 50: number analyzed (Participants) | 41
  Week 8: PASI 50 | 82.9
  Week 12: PASI 100 | 34.1
  Week 12: PASI 90 | 63.6
  Week 12: PASI 75 | 84.1
  Week 12: PASI 50 | 93.2
  Week 16: PASI 100: number analyzed (Participants) | 42
  Week 16: PASI 100 | 40.5
  Week 16: PASI 90: number analyzed (Participants) | 42
  Week 16: PASI 90 | 66.7
  Week 16: PASI 75: number analyzed (Participants) | 42
  Week 16: PASI 75 | 83.3
  Week 16: PASI 50: number analyzed (Participants) | 42
  Week 16: PASI 50 | 97.6
  Week 28: PASI 100: number analyzed (Participants) | 42
  Week 28: PASI 100 | 38.1
  Week 28: PASI 90: number analyzed (Participants) | 42
  Week 28: PASI 90 | 81.0
  Week 28: PASI 75: number analyzed (Participants) | 42
  Week 28: PASI 75 | 92.9
  Week 28: PASI 50: number analyzed (Participants) | 42
  Week 28: PASI 50 | 92.9
  Week 40: PASI 100: number analyzed (Participants) | 42
  Week 40: PASI 100 | 42.9
  Week 40: PASI 90: number analyzed (Participants) | 42
  Week 40: PASI 90 | 78.6
  Week 40: PASI 75: number analyzed (Participants) | 42
  Week 40: PASI 75 | 90.5
  Week 40: PASI 50: number analyzed (Participants) | 42
  Week 40: PASI 50 | 92.9
  Week 52: PASI 100: number analyzed (Participants) | 41
  Week 52: PASI 100 | 53.7
  Week 52: PASI 90: number analyzed (Participants) | 41
  Week 52: PASI 90 | 70.7
  Week 52: PASI 75: number analyzed (Participants) | 41
  Week 52: PASI 75 | 87.8
  Week 52: PASI 50: number analyzed (Participants) | 41
  Week 52: PASI 50 | 92.7

7. Secondary Outcome: Percent Change From Baseline in PASI Score at Weeks 4, 8, 12, 16, 28, 40, and 52
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72 (disease severity). PASI 100 responders were defined as 100% improvement in PASI from Baseline respectively. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 28, 40, 52
Population: FAS. For participants meeting one or more TF criteria, were considered to have 0% improvement from baseline. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
percent change
  Week 4: number analyzed (Participants) | 42
  Week 4 | 52.9 (27.33)
  Week 8: number analyzed (Participants) | 41
  Week 8 | 78.9 (21.44)
  Week 12: number analyzed (Participants) | 42
  Week 12 | 89.7 (13.80)
  Week 16: number analyzed (Participants) | 42
  Week 16 | 90.4 (13.77)
  Week 28: number analyzed (Participants) | 42
  Week 28 | 90.4 (21.55)
  Week 40: number analyzed (Participants) | 42
  Week 40 | 89.9 (23.01)
  Week 52: number analyzed (Participants) | 41
  Week 52 | 89.1 (24.28)

8. Secondary Outcome: Percentage of Participants Who Achieved PASI 100, PASI 90, PASI 75 or PASI 50 Response in PASI Components (Induration, Erythema, and Scaling) and Region Components (Head, Trunk, Upper Extremities, and Lower Extremities) at Week 12
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90 percentage (%)-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72 (disease severity). PASI 50, 75, 90, and 100 responders were defined as >=50%, >=75%, >=90%, and 100% improvement in PASI component from Baseline respectively. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Week 12
Population: FAS. Participants meeting one or more TF criteria were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
percentage of participants
  Induration: PASI 100 | 43.2
  Induration: PASI 90 | 61.4
  Induration: PASI 75 | 77.3
  Induration: PASI 50 | 93.2
  Scaling: PASI 100 | 38.6
  Scaling: PASI 90 | 63.6
  Scaling: PASI 75 | 84.1
  Scaling: PASI 50 | 90.9
  Erythema: PASI 100 | 38.6
  Erythema: PASI 90 | 61.4
  Erythema: PASI 75 | 81.8
  Erythema: PASI 50 | 93.2
  Head: PASI 100 | 52.3
  Head: PASI 90 | 65.9
  Head: PASI 75 | 79.5
  Head: PASI 50 | 93.2
  Trunk: PASI 100 | 61.4
  Trunk: PASI 90 | 61.4
  Trunk: PASI 75 | 79.5
  Trunk: PASI 50 | 88.6
  Upper extremities: PASI 100 | 65.9
  Upper extremities: PASI 90 | 65.9
  Upper extremities: PASI 75 | 79.5
  Upper extremities: PASI 50 | 84.1
  Lower extremities: PASI 100 | 68.2
  Lower extremities: PASI 90 | 68.2
  Lower extremities: PASI 75 | 72.7
  Lower extremities: PASI 50 | 93.2

9. Secondary Outcome: Change From Baseline in Children Dermatology Life Quality Index (CDLQI) Score at Weeks 4, 12, 28, and 52
Description: CDLQI was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (Not at all) to 3 (Very much). The total score ranges from 0 to 30. The higher the score, the greater the impairment in quality of life (QoL). TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Baseline and Weeks 4, 12, 28, 52
Population: FAS. Participants who met TF criteria prior to Week 12 were assigned 0 change. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 44
units on a scale
  Week 4: number analyzed (Participants) | 42
  Week 4 | -4.1 (4.88)
  Week 12: number analyzed (Participants) | 42
  Week 12 | -6.3 (6.43)
  Week 28: number analyzed (Participants) | 42
  Week 28 | -6.6 (5.79)
  Week 52: number analyzed (Participants) | 41
  Week 52 | -6.4 (6.10)

10. Secondary Outcome: Percentage of Participants With a CDLQI Score of 0 or 1 at Week 12 in Participants With a Baseline CDLQI Score Greater Than (>) 1
Description: CDLQI was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (Not at all) to 3 (Very much). The total score ranges from 0 to 30. The higher the score, the greater impairment in quality of life. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Week 12
Population: FAS with CDLQI score > 1 at baseline. Participants who met 1 or more TF criteria prior to Week 12 or with missing data were considered as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 39
percentage of participants | 61.5 [44.6 to 76.6]

11. Secondary Outcome: Percentage of Participants With a CDLQI Score of 0 or 1 at Weeks 4, 12, 28 and 52 in Participants With a Baseline CDLQI Score > 1
Description: CDLQI was used to assess the impact of psoriasis on subject health-related quality of life. The CDLQI has 10 items assessing health-related quality of life (HRQOL) in patients with skin disease each measured on a scale from 0 (Not at all) to 3 (Very much). The total score ranges from 0 to 30. The total score ranges from 0 to 30. The higher the score, the greater impairment in quality of life. TF criteria- discontinued study agent due to lack of efficacy or adverse event of psoriasis or who started protocol-prohibited medication/therapy.
Time Frame: Weeks 4, 12, 28, and 52
Population: FAS with CDLQI > 1 at baseline. Participants who met 1 or more TF criteria were considered as nonresponders after TF. In addition, participants with missing data at Week 12 were considered as nonresponders at Week 12. Here 'n' (number analyzed) included all participants who were evaluable at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 39
percentage of participants
  Week 4: number analyzed (Participants) | 37
  Week 4 | 37.8
  Week 12 | 61.5
  Week 28: number analyzed (Participants) | 37
  Week 28 | 62.2
  Week 52: number analyzed (Participants) | 36
  Week 52 | 58.3

12. Secondary Outcome: Change From Baseline in CDLQI Component Scores at Week 12
Description: as for outcome 11
Time Frame: Baseline and Week 12
Population: FAS. Participants who met TF criteria prior to Week 12 were assigned 0 change. Here 'N' (number of participants analyzed) included all participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ustekinumab Standard Dosage (Main Study)
Number analyzed (Participants) | 42
units on a scale
  Symptoms and feelings | -1.9 (1.81)
  Leisure | -1.7 (2.19)
  School or holidays | -0.5 (0.80)
  Personal relationships | -0.8 (1.71)
  Sleep | -0.4 (0.91)
  Treatment | -0.9 (1.14)

13. Secondary Outcome: Percentage of Participants With PGA Score of Cleared (0), Cleared (0) or Minimal (1), Cleared (0) or Minimal (1) or Mild (2) at Weeks 80, 104, 128, 152, and 176
Description: The PGA is used to determine the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), marked (4), or severe (5). Higher scores indicated worse disease.
Time Frame: Weeks 80, 104, 128, 152, 176
Population: FAS; all participants enrolled in the LTE who received at least an injection of ustekinumab at Week 56 (partial or complete). Here "N" (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed): participants evaluated at given timepoints.
Measure: Number; unit: percentage of participants
Groups:
- Ustekinumab Standard Dosage (Long-Term Extension [LTE]): Participants who had a beneficial response from ustekinumab treatment continued receiving ustekinumab weight based dose in a every 12 weeks (q12w) regimen from Week 56 onwards until commercially available or marketing authorization being denied or up to Week 264. Ustekinumab was administered as SC injections of 0.75 mg/kg for participants with weight <60 kg, 45 mg for participants with weight >=60 kg to <=100 kg, and 90 mg for participants with weight >100 kg.
Arm/Group | Ustekinumab Standard Dosage (Long-Term Extension [LTE])
Number analyzed (Participants) | 25
percentage of participants
  Week 80: PGA score 0 | 64
  Week 80: PGA score 0 or 1 | 80
  Week 80: PGA score 0 or 1 or 2 | 100
  Week 104: PGA score 0: number analyzed (Participants) | 20
  Week 104: PGA score 0 | 50
  Week 104: PGA score 0 or 1: number analyzed (Participants) | 20
  Week 104: PGA score 0 or 1 | 70
  Week 104: PGA score 0 or 1 or 2: number analyzed (Participants) | 20
  Week 104: PGA score 0 or 1 or 2 | 100
  Week 128: PGA score 0: number analyzed (Participants) | 20
  Week 128: PGA score 0 | 60
  Week 128: PGA score 0 or 1: number analyzed (Participants) | 20
  Week 128: PGA score 0 or 1 | 80
  Week 128: PGA score 0 or 1 or 2: number analyzed (Participants) | 20
  Week 128: PGA score 0 or 1 or 2 | 95
  Week 152: PGA score 0: number analyzed (Participants) | 13
  Week 152: PGA score 0 | 53.8
  Week 152: PGA score 0 or 1: number analyzed (Participants) | 13
  Week 152: PGA score 0 or 1 | 61.5
  Week 152: PGA score 0 or 1 or 2: number analyzed (Participants) | 13
  Week 152: PGA score 0 or 1 or 2 | 100
  Week 176: PGA score 0: number analyzed (Participants) | 3
  Week 176: PGA score 0 | 33.3
  Week 176: PGA score 0 or 1: number analyzed (Participants) | 3
  Week 176: PGA score 0 or 1 | 66.7
  Week 176: PGA score 0 or 1 or 2: number analyzed (Participants) | 3
  Week 176: PGA score 0 or 1 or 2 | 100

ADVERSE EVENTS:
Time Frame: Up to Week 264
Description: The safety analysis set included all the enrolled participants who received at least 1 injection of ustekinumab (partial or complete) during the study.
Groups:
- Ustekinumab Standard Dosage (Main Study): Participants received ustekinumab standard weight-based dose at Weeks 0 and 4 followed by every 12 weeks (q12w) dosing up to Week 40. Ustekinumab was administered as subcutaneous (SC) injections of 0.75 milligrams per kilogram (mg/kg) for participants with weight less than (<) 60 kilograms (kg), 45 mg for participants with weight greater than or equal to (>=) 60 kg to less than or equal to (<=) 100 kg, and 90 mg for participants with weight > 100 kg. Participants had a safety follow-up till Week 56.
Arm/Group | Ustekinumab Standard Dosage (Main Study) | Ustekinumab Standard Dosage (Long-Term Extension [LTE])
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/28
Serious Adverse Events (participants affected / at risk) | 3/44 | 1/28
Other Adverse Events (participants affected / at risk) | 27/44 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab Standard Dosage (Main Study) (N=44) | Ustekinumab Standard Dosage (Long-Term Extension [LTE]) (N=28)
Infectious Mononucleosis (Infections and infestations) | 1 | 0
Eyelid Injury (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab Standard Dosage (Main Study) (N=44) | Ustekinumab Standard Dosage (Long-Term Extension [LTE]) (N=28)
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Injection Site Erythema (General disorders) | 6 | 2
Gastroenteritis (Infections and infestations) | 3 | 3
Nasopharyngitis (Infections and infestations) | 11 | 8
Otitis Media (Infections and infestations) | 3 | 2
Pharyngitis (Infections and infestations) | 6 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 4 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Due to the study design, the population was limited in the long-term extension period and decreased over time as participants met discontinuation criteria and exited the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT02698475/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02698475/SAP_001.pdf